CLINICAL TRIAL: NCT03628352
Title: An Open-Label Taste Assessment of Tricaprilin Formulated as a Powder for Reconstitution in Healthy Panelists
Brief Title: Taste-masking Study for Tricaprilin in Sensory Panelists
Acronym: TMS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AC-18-019_TM
Record Dates: First submitted 2018-08-08; First posted 2018-08-14 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Taste Profile Assessments
MeSH Terms: interventions — tricaprylin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tricaprilin (Experimental): Approximately 5 mL liquid of tricaprilin using various flavoring agents (swish and expectorate) up to 20 times. Dose will not be ingested.
  Interventions: Drug: Tricaprilin

INTERVENTIONS:
Drug: Tricaprilin — Tricaprilin with flavoring agents added

SUMMARY:
This is an open-label multiple-dose study of the taste profile of tricaprilin formulated as a powder for reconstitution.

ELIGIBILITY:
Inclusion Criteria:

1. The healthy male or female sensory panelist is between 25 and 80 years of age (inclusive) who volunteers for study participation and is able to read, understand, and sign and date a written informed consent form (ICF) before study participation.
2. The panelist is male, or is a non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol, or is a female of non-childbearing potential.
3. The sensory panelist is qualified based on training and experience.
4. The panelist is able to perform the required procedures according to the specified methodology
5. The panelist has provided full written consent to participate in the study.

Exclusion Criteria:

1. The sensory panelist has a history of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug(s) to the sensory panelist.
2. The sensory panelist has a known sensitivity to medium-chain triglycerides (MCTs) or any of the excipients used in study formulations.
3. The sensory panelist has a known history of kidney disease, inflammatory bowel disease, or Bradycardia. .
4. If female, the sensory panelist is pregnant, nursing, planning to become pregnant during the study.
5. Panelist must not have any planned hospitalizations or in-patient surgical procedures that are scheduled to take place during the study.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Taste as assessed by trained sensory panelists | 1 day
  single dose (swish and expectorate)
Smell as assessed by trained sensory panelists | 1 day
Texture as assessed by trained sensory panelists | 1 day
  single dose (swish and expectorate)
Palatability as assessed by trained sensory panelists | 1 day
  single dose (swish and expectorate)

CONTACTS AND LOCATIONS:
Overall Officials: Carol McKenna, Principal Investigator — Senopsys
Locations (1):
- Senopsys, Inc., Woburn, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No